CLINICAL TRIAL: NCT05213767
Title: Phase I Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB2916 Injection in Patients With Advanced Malignant Tumors
Brief Title: Clinical Study to Evaluate the Tolerability and Pharmacokinetics of TQB2916 Injection in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2916- I -01
Record Dates: First submitted 2022-01-26; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2916 injection (Experimental): 2.5mg/ quaque die (QD) was used as the initial dose, 21 days as a treatment cycle. The drug is administered on the first day of each cycle until the disease progresses or the investigator judges that it is not suitable for subject to continue to take medicine.
  Interventions: Drug: TQB2916 injection

INTERVENTIONS:
Drug: TQB2916 injection — TQB2916 injection is a kind of Tumor necrosis factor receptor superfamily member 5 (CD40) agonist, which is a humanized immunoglobulinG2 (IgG2) monoclonal antibody targeting CD40. This product can bind to CD40 on target cells to activate downstream signaling pathways and generate anti-tumor immune responses. At the same time, it can promote the apoptosis of B-cell lymphoma Ramos cells.

SUMMARY:
This project is an open, dose escalation and expansion phase I clinical study. The first phase is a dose escalation study, and the second phase is a dose expansion study based on the Maximum tolerated dose (MTD) / Recommended Phase II Dose (RP2D) obtained in the first phase. The purpose is to evaluate the safety, tolerability, and pharmacokinetic characteristics of TQB2916 injection in patients with advanced tumors, and to initially evaluate the antitumor efficacy of TQB2916 injection.

ELIGIBILITY:
Inclusion Criteria:

* 1 Subjects with advanced malignant tumors clearly diagnosed by pathology and / or cytology, lack of conventional effective treatment methods, failure or relapse after treatment.
* 2 18-75 years old; Eastern Cooperative Oncology Group (ECOG) physical status: 0-1; at least 3 months expected survival period.
* 3 The function of main organs is normal.
* 4 Subjects must need to adopt effective methods of contraception.
* 5 Subjects voluntarily joined the study, signed informed consent form, and with good compliance.

Exclusion Criteria:

* 1 Patients has had or is currently having other malignant tumors within 3 years. The following two conditions can be included in the group: other malignant tumors treated with a single operation to achieved R0 resection without recurrence and metastasis. Cured cervical carcinoma in situ, non-melanoma skin cancer, nasopharyngeal carcinoma and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)].
* 2 The toxicity of previous antitumor treatment is not recovered to ≤ grade 1 (Common Terminology Criteria for Adverse Events (CTCAE) 5.0).
* 3 Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before treatment.
* 4 Subjects had an arteriovenous thrombosis event within 6 months.
* 5 Subjects occurred Evans syndrome within 3 months.
* 6 History of drug abuse, alcohol or drug abuse or mental disorder.
* 7 Subjects who suffered from Active tuberculosis within 1 year.
* 8 The subjects had any history of bleeding or coagulopathy.
* 9 Cirrhosis, active hepatitis.
* 10 The subjects was diagnosed with renal failure and required hemodialysis or peritoneal dialysis.
* 11 History of immunodeficiency, including positive human immunodeficiency virus (HIV) test or other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* 12 Subjects who have epilepsy and require treatment.
* 13 Received the treatment of proprietary Chinese medicines with anti-tumor indications clearly stated in the National Medical Products Administration (NMPA) approved drug instructions within 2 weeks of starting treatment.
* 14 The symptoms of subjects with known central nervous system metastasis, spinal cord compression, meningeal metastasis, or leptomeningeal disease.
* 15 Vaccination history of live attenuated vaccine before 28 days of starting treatment, or planned vaccination of live attenuated vaccine during the study period.
* 16 History of severe allergy to macromolecule drugs or known components of TQB2916 injection.
* 17 Receiving any other investigational agent within 4 weeks before first dose.
* 18 According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 52 weeks
  To evaluate MTD of TQB2916 injection in patients with advanced solid tumors
Dose limited toxicity (DLT) | Baseline up to 52 weeks
  To evaluate DLT of TQB2916 injection in Chinese adult patients with advanced solid tumors
Recommended Phase II Dose (RP2D) | Baseline up to 52 weeks
  To evaluate RP2D of TQB2916 injection in Chinese adult patients with advanced solid tumors

SECONDARY OUTCOMES:
Adverse events (AE) , serious adverse events (SAE) and treatment-related adverse events (TRAE) | Baseline up to 104 weeks
  The occurrence of all adverse events (AE), serious adverse events (SAE) and treatment-related adverse events (TRAE)
Tmax | (-1 to 0 hour) (pre-dose), 0，1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  Time to reach maximum (peak) plasma concentration following drug administration
Maximum (peak) plasma drug concentration (Cmax) | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  Cmax is the maximum plasma concentration of TQB2916.
Elimination half-life (t1/2) | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  t1/2 is time it takes for the blood concentration of TQB2916 or metabolite(s) to drop by half.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  To characterize the pharmacokinetics of TQB2916 by assessment of area under the plasma concentration time curve from the first dose to infinity.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  Cmax is the maximum plasma concentration of TQB2916
Concentration at the end of the dosing interval AUCtau,ss | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  To characterize the pharmacokinetics of TQB2916 by assessment of area The concentration at the end of the administration interval
Minimum steady-state plasma drug concentration during a dosage interval (Css-min) | (-1 to 0 hour) (pre-dose), 0, 1, 2, 4, 8, 24, 48,72,144,312,480 hours after intravenous injection of Cycle 1/3 Day 1; In 1 hour before intravenous injection on Cycle 2 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, Cycle 7 Day 1 and Cycle 8 Day 1.
  Cmin is the minimum plasma concentration of TQB2916
Progress Free Survival (PFS) | up to 96 weeks
  Time from the first dose to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Disease control rate (DCR) | up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 96 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Overall survival (OS) | up to 96 weeks
  the time from start of study treatment to date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China